CLINICAL TRIAL: NCT04050605
Title: Refitting Somofilcon A Toric Contact Lens Wearers Into Fanfilcon A Toric Lenses for 4-weeks of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EX-MKTG-102
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2020-08-28 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: First pair of study lenses (habitual lenses - somofilcon A toric) will be dispensed and worn for 4-weeks of daily wear, then second pair of lenses (test lenses - fanfilcon A toric) will be dispensed and worn for 4-weeks for daily wear.
Masking Description: Study lenses will be transferred, by an assistant, out of their packaging to unmarked new contact lens cases filled with preservative free sterile saline just prior to dispensing to maintain subject masking of the study lenses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- somofilcon A toric (habitual), then fanfilcon toric (test) (Experimental): Participants are habitual wearers of somofilcon A toric lens and refitted with fanfilcon A toric lens.
  Interventions: Device: somofilcon A toric contact lens; Device: fanfilcon A toric contact lens

INTERVENTIONS:
Device: somofilcon A toric contact lens — Contact Lens
  Other Names: Habitual lens
Device: fanfilcon A toric contact lens — Contact Lens
  Other Names: Test Lens

SUMMARY:
The aim of this prospective study is to evaluate the clinical performance of habitual wearers of Clariti Toric lenses after a refit with Avaira Vitality Toric lenses for 1-month of daily wear.

DETAILED DESCRIPTION:
The aim of this prospective study is to evaluate the clinical performance of habitual wearers of Clariti Toric lenses after a refit with Avaira Vitality Toric lenses for 1-month of daily wear.

This is a prospective, subject masked; bilateral, 1-month refit study comparing the fitting characteristics of Clariti Toric silicone hydrogel lenses, (somofilcon A); against Avaira Vitality silicone hydrogel Toric lenses (fanfilcon A).

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft toric contact lens wearer
* Has a contact lens spherical prescription between +6.00 to -8.00 (inclusive)
* Have no less than -0.75D of astigmatism and no more than -2.25 D in both eyes.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Patient contact lens refraction should fit within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has a CL prescription outside the range of the available parameters of the study lenses.
* Has a spectacle cylinder less than -0.75D or more than -2.50 D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 (0.10 logMAR) in either eye.
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:
* Pathological dry eye or associated findings
* Pterygium, pinguecula, or corneal scars within the visual axis
* Neovascularization > 0.75 mm in from of the limbus
* Giant papillary conjunctivitis (GCP) worse than grade 1
* Anterior uveitis or iritis (past or present)
* Seborrheic eczema, Seborrheic conjunctivitis
* History of corneal ulcers or fungal infections
* Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has Presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Velázquez Guerrero, MSc., FIACLE, Principal Investigator — School of Optometry, National Autonomous University (UNAM), Mexico City
Locations (1):
- Optometry Clinic, National Autonomous University, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Somofilcon A Toric (Habitual), Then Fanfilcon Toric (Test)
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Somofilcon A Toric (Habitual), Then Fanfilcon Toric (Test)
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mexico | 40

OUTCOME MEASURES:

1. Primary Outcome: Lens Centration - Somofilcon A Toric (Habitual) Lens
Description: Lens Centration assessed using a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Groups:
- Somofilcon A Toric (Habitual): Participants wore their habitual somofilcon A toric lens for 4-weeks.
  somofilcon A toric contact lens: Contact Lens
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
percentage of lenses
  Optimum | 100
  Acceptable | 0
  Unacceptable | 0

2. Primary Outcome: Lens Centration - Somofilcon A Toric (Habitual) Lens
Description: Lens Centration (using a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: 4 weeks
Measure: Number; unit: percentage of lenses
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
percentage of lenses
  Optimum | 100
  Acceptable | 0
  Unacceptable | 0

3. Primary Outcome: Lens Centration - Fanfilcon A Toric Lens
Description: Lens Centration using a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Groups:
- Fanfilcon A Toric Lens: Participants were refitted with fanfilcon A toric lens.
  fanfilcon A toric contact lens: Contact Lens
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
percentage of lenses
  Optimum | 100
  Acceptable | 0
  Unacceptable | 0

4. Primary Outcome: Lens Centration - Fanfilcon A Toric Lens
Description: Lens Centration using a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: 2-weeks
Measure: Number; unit: percentage of lenses
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
percentage of lenses
  Optimum | 100
  Acceptable | 0
  Unacceptable | 0

5. Primary Outcome: Lens Centration - Fanfilcon A Toric Lens
Description: Lens Centration using a 3-point scale (1=optimal centration, 2=decentration acceptable, 3=decentration unacceptable).
Time Frame: 4-weeks
Measure: Number; unit: percentage of lenses
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
percentage of lenses
  Optimum | 100
  Acceptable | 0
  Unacceptable | 0

6. Primary Outcome: Corneal Coverage - Somofilcon A Toric (Habitual ) Lens
Description: Corneal Coverage (Yes = full corneal coverage all time / no= incomplete corneal coverage)
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
percentage of lenses
  Yes | 100
  No | 0

7. Primary Outcome: Corneal Coverage - Somofilcon A Toric (Habitual ) Lens
Description: Corneal Coverage (Yes = full corneal coverage all time / no= incomplete corneal coverage)
Time Frame: 4-weeks
Measure: Number; unit: percentage of lenses
Groups:
- Somofilcon A Toric (Habitual): Participants wore their habitual somofilcon A toric lens for 4-weeks..
  somofilcon A toric contact lens: Contact Lens
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
percentage of lenses
  Yes | 100
  No | 0

8. Primary Outcome: Corneal Coverage - Fanfilcon A Toric Lens
Description: Corneal Coverage (Yes = full corneal coverage all time / no= incomplete corneal coverage)
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
percentage of lenses
  Yes | 100
  No | 0

9. Primary Outcome: Corneal Coverage - Fanfilcon A Toric Lens
Description: Corneal Coverage (Yes = full corneal coverage all time / no= incomplete corneal coverage)
Time Frame: 2-weeks
Measure: Number; unit: percentage of lenses
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
percentage of lenses
  Yes | 100
  No | 0

10. Primary Outcome: Corneal Coverage - Fanfilcon A Toric Lens
Description: Corneal Coverage (Yes = full corneal coverage all time / no= incomplete corneal coverage)
Time Frame: 4-weeks
Measure: Number; unit: percentage of lenses
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
percentage of lenses
  Yes | 100
  No | 0

11. Primary Outcome: Post-Blink Movement - Somofilcon A Toric (Habitual) Lens
Description: Post-Blink movement (0-4 Scale, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
units on a scale | 2.0 (0.0)

12. Primary Outcome: Post-Blink Movement - Somofilcon A Toric (Habitual) Lens
Description: as for outcome 11
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Somofilcon A Toric (Habitual): Participants wore their habitual somofilcon A toric lens for 4 weeks.
  somofilcon A toric contact lens: Contact Lens
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
units on a scale | 2.0 (0.0)

13. Primary Outcome: Post-Blink Movement - Fanfilcon A Toric Lens
Description: as for outcome 11
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
units on a scale | 2.0 (0.0)

14. Primary Outcome: Post-Blink Movement - Fanfilcon A Toric Lens
Description: as for outcome 11
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
units on a scale | 2.0 (0.0)

15. Primary Outcome: Post-Blink Movement - Fanfilcon A Toric Lens
Description: Post-Blink movement (0-4 Scale,0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement).
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A Toric Lens
Number analyzed (Participants) | 40
units on a scale | 2.0 (0.0)

16. Primary Outcome: Overall Lens Fit Acceptance - Somofilcon A Toric (Habitual) Lens
Description: Overall fit acceptance - using a 0 - 4 scale (where 0 = should not be worn, 1 = borderline but unacceptable, 2 = min. acceptable, early review, 3 = not perfect but OK to dispense, and 4 = perfect).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
units on a scale | 3.8 (0.5)

17. Primary Outcome: Overall Lens Fit Acceptance - Somofilcon A Toric (Habitual) Lens
Description: as for outcome 16
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
units on a scale | 3.8 (0.5)

18. Primary Outcome: Overall Lens Fit Acceptance - Fanfilcon A Toric Lens
Description: as for outcome 16
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- fanfilconA Toric: Participants were their refitted with fanfilcon A toric lens for 4-weeks..
  fanfilcon A toric contact lens: Contact Lens
Arm/Group | fanfilconA Toric
Number analyzed (Participants) | 40
units on a scale | 3.9 (0.3)

19. Primary Outcome: Overall Lens Fit Acceptance - Fanfilcon A Toric Lens
Description: as for outcome 16
Time Frame: 2-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | fanfilconA Toric
Number analyzed (Participants) | 40
units on a scale | 4.0 (0.2)

20. Primary Outcome: Overall Lens Fit Acceptance - Fanfilcon A Toric Lens
Description: as for outcome 16
Time Frame: 4-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | fanfilconA Toric
Number analyzed (Participants) | 40
units on a scale | 4.0 (0.2)

21. Secondary Outcome: Average Daily Wearing Time - Somofilcon A Toric (Habitual) Lens
Description: Average Daily Wearing Time for somofilcon A toric (habitual) lens measured by hours/day.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
hours/day | 10.4 (3.0)

22. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A Toric Lens
Description: Average Daily Wearing Time for fanfilcon A toric lens measured by hours/day.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Groups:
- Fanfilcon A Toric: Participants were refitted with fanfilcon A toric lens for 4-weeks..
  fanfilcon A toric contact lens: Contact Lens
Arm/Group | Fanfilcon A Toric
Number analyzed (Participants) | 40
hours/day | 10.5 (2.7)

23. Secondary Outcome: Average Daily Wearing Time - Fanfilcon A Toric Lens
Description: Average Daily Wearing Time for fanfilcon A toric lens measured by hours/day.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A Toric
Number analyzed (Participants) | 40
hours/day | 10.9 (2.6)

24. Secondary Outcome: Average Comfortable Wearing Time - Somofilcon A Toric (Habitual) Lens
Description: Average Comfortable Wearing Time - somofilcon A toric (habitual) lens measured by hours/day
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Somofilcon A Toric (Habitual)
Number analyzed (Participants) | 40
hours/day | 8.4 (3.5)

25. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A Toric Lens
Description: Average comfortable Wearing Time for fanfilcon A toric lens measured by hours/day.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A Toric
Number analyzed (Participants) | 40
hours/day | 9.0 (2.6)

26. Secondary Outcome: Average Comfortable Wearing Time - Fanfilcon A Toric Lens
Description: Average comfortable Wearing Time for fanfilcon A toric lens measured by hours/day.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Fanfilcon A Toric
Number analyzed (Participants) | 40
hours/day | 9.6 (2.6)

ADVERSE EVENTS:
Time Frame: From dispense up to 4-weeks for each lens type, a total of 8-weeks.
Groups:
- Somofilcon A Toric (Habitual) Lens: Participants are habitual wearers of somofilcon A toric lens for 4-weeks
  somofilcon A toric contact lens: Contact Lens
- Fanfilcon A Toric Contact Lens: Participants were refitted with fanfilcon A toric lens for 4-weeks
  fanfilcon A toric contact lens: Contact Lens
Arm/Group | Somofilcon A Toric (Habitual) Lens | Fanfilcon A Toric Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT04050605/Prot_SAP_000.pdf